CLINICAL TRIAL: NCT00400075
Title: CHUSPAN PAN BP Treatment of Polyarteritis Nodosa and Microscopic Polyangiitis Without Poor-Prognosis Factors a Prospective Randomized Study in 125 Patients
Brief Title: CHUSPAN PAN BP Treatment of Polyarteritis Nodosa and Microscopic Polyangiitis Without Poor-Prognosis Factors
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 95.067/2
Record Dates: First submitted 2006-11-14; First posted 2006-11-16 (Estimated); Last update posted 2006-11-16 (Estimated); Status verified 2006-11

CONDITIONS: Polyarteritis Nodosa; Microscopic Polyangiitis
Keywords: Polyarteritis; Vasculitis; Therapy; Cyclophosphamide; Azathioprine
MeSH Terms: conditions — Polyarteritis Nodosa; Microscopic Polyangiitis; Vasculitis | interventions — Azathioprine; Cyclophosphamide

INTERVENTIONS:
Drug: azathioprine
Drug: cyclophosphamide

SUMMARY:
To assess the efficacy of systemic corticosteroids alone as first-line treatment of polyarteritis nodosa and microscopic polyangiitis without poor-prognosis factors as defined by the five-factor score (FFS=0), and to compare the efficacy and safety of azathioprine vs pulse cyclophosphamide as adjunctive immunosuppressive therapy to treat failure or relapse.

DETAILED DESCRIPTION:
All patients initially treated with systemic corticosteroids alone: optional IV methylprednisolone pulse (15 mg/kg) at treatment start followed by oral prednisone (1 mg/kg/day) according to a tapering schedule. Treating physicians allowed to treat minor relapses with corticosteroids without referring the patient for randomization, as long as the prednisone dose did not exceed 0.5 mg/kg for 1 month.

Patients in whom prednisone doses could not be tapered below 20 mg, those who failed to enter remission and those who relapsed were randomized to receive either 6 months of oral azathioprine (2mg/kg/day) or 6 cyclophosphamide pulses (0.6g/m2 D1, D15, D30 then every month)

ELIGIBILITY:
Inclusion Criteria:

* Men and women with newly diagnosed polyarteritis nodosa or microscopic polyangiitis;
* absence of poor prognostic factors as defined by the five-factor score (serum creatinine > 140 μmol/l or 1.58 mg/dl, proteinuria > 1 g/day, severe gastrointestinal tract involvement, specific cardiomyopathy and/or central nervous system involvement;
* written informed consent.
* Both genders eligible;
* age ≥ 15 years.

Exclusion Criteria:

* age < 15 years, previously treated systemic vasculitis;
* history of cancer;
* pregnant or breast-feeding women;
* psychiatric disorders that might compromise compliance with therapy;
* contraindication to study drug;
* other ongoing therapeutic trial;
* concomitant viral hepatitis B or C or human immunodeficiency virus (HIV) infection

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124
Dates: Start 1996-07

PRIMARY OUTCOMES:
Number of events (failures, relapses and/or deaths) occurring in each group, defining the disease-free survival rate, measured at study end (mean follow-up of 5 years)

SECONDARY OUTCOMES:
Overall survival, relapse rate and adverse events, measured at study end (mean follow-up of 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Cordier, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Camillo Ribi, Geneva, Switzerland

REFERENCES:
- [Derived] Samson M, Puechal X, Devilliers H, Ribi C, Cohen P, Bienvenu B, Terrier B, Pagnoux C, Mouthon L, Guillevin L; French Vasculitis Study Group (FVSG). Mononeuritis multiplex predicts the need for immunosuppressive or immunomodulatory drugs for EGPA, PAN and MPA patients without poor-prognosis factors. Autoimmun Rev. 2014 Sep;13(9):945-53. doi: 10.1016/j.autrev.2014.08.002. Epub 2014 Aug 19. PMID 25153486